CLINICAL TRIAL: NCT04064658
Title: Effects of Remote Ischemic Pre-Conditioning on Neurologic Complications in Adult Ischemic Moyamoya Disease Patients Undergoing Encephaloduroarteriosynangiosis
Brief Title: Effects of Remote Ischemic Pre-Conditioning in Moyamoya Disease Patients
Acronym: RIME
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: waiting for the ethics approval of collaborator affiliation
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Peking University International Hospital (Other)
Responsible Party: Principal Investigator, yuanli Zhao, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIPC2019
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-07

CONDITIONS: Moyamoya Disease; Remote Ischemic Preconditioning
Keywords: Moyamoya Disease; Cerebrovascular Disorders; Arterial Occlusive Diseases; Ischemia
MeSH Terms: conditions — Moyamoya Disease; Cerebrovascular Disorders; Arterial Occlusive Diseases; Ischemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham RIPC group (Sham Comparator): Treatment:Patients in this group received standard medical therapy and sham remote ischemic preconditioning treatment.
  Device:Sham RIPC consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by a sphygmomanometer placed on bilateral arm and inflated to 60 mmHg for 5-min followed by deflating the cuff for 5-min, each patient in Sham RIPC group do it twice a day for at least five days before encephaloduroarteriosynangiosis.
  Procedure: Encephaloduroarteriosynangiosis
  Interventions: Procedure: Sham remote ischemic preconditioning; Procedure: Encephaloduroarteriosynangiosis
- RIPC group (Experimental): Treatment:Patients in this group received standard medical therapy and remote ischemic preconditioning (RIPC) treatment.
  Device:RIPC consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by a sphygmomanometer placed on bilateral arm and inflated to 200 mmHg for 5-min followed by deflating the cuff for 5-min,each patient in the RIPC group do it twice a day for at least five days before encephaloduroarteriosynangiosis.
  Procedure: Encephaloduroarteriosynangiosis
  Interventions: Procedure: Remote ischemic preconditioning; Procedure: Encephaloduroarteriosynangiosis

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Remote ischemic preconditioning consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by a sphygmomanometer placed on bilateral arm and inflated to 200 mmHg for 5-min followed by deflating the cuff for 5-min.
  Other Names: RIPC
  Arms: RIPC group
Procedure: Sham remote ischemic preconditioning — Sham remote ischemic preconditioning consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, which is induced by a sphygmomanometer placed on bilateral arm and inflated to 60 mmHg for 5-min followed by deflating the cuff for 5-min.
  Other Names: Sham RIPC
  Arms: Sham RIPC group
Procedure: Encephaloduroarteriosynangiosis — Encephaloduroarteriosynangiosis is an indirect revascularization surgery of moyamoya disease
  Other Names: EDAS

SUMMARY:
In the present study, investigators evaluated whether RIPC reduce the major neurological complications in adult moyamoya disease patients undergoing encephaloduroarteriosynangiosis (EDAS).

DETAILED DESCRIPTION:
BACKGROUND: Brain ischemia and injury contributed to perioperative morbidity and mortality in revascularization surgery. Remote ischemic preconditioning (RIPC), brief periods of ischemia followed by reperfusion, can provide systemic protection for prolonged ischemia. Previous study found combined remote ischemic pre- and post-conditioning can be effective in reducing neurologic complications and the duration of hospitalization in moyamoya patients undergoing direct revascularization.In order to investigate whether RIPC before EDAS can protect these patients from the perioperative and long-term complications, a prospective randomized controlled trial will be performed in the current study.

DESIGNING: About 328 patients who are eligible for carotid artery stenting will be randomly assigned in 1:1 ratio to RIPC group and sham RIPC group (control). Remote limb ischemic preconditioning (RIPC) is consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, it is induced by a sphygmomanometer placed on bilateral arm and inflated to 200 mmHg for 5-min followed by deflating the cuff for 5-min, patients in the RIPC group will do it twice a day for at least five days before EDAS. Patients in the sham RIPC group receive sham RIPC treatment, which is consisted of five 5-min cycles of bilateral arm ischemia/reperfusion, induced by a sphygmomanometer placed on bilateral arm and inflated to 60 mmHg for 5-min followed by deflating the cuff for 5-min, they will do it twice a day for at least five days before EDAS. Cerebral injury is assessed by plasma Human Soluble protein-100B (S-100B) and Neuron specific enolase (NSE). Clinical outcomes are determined by cerebrovascular events (including ischemic stroke, transient ischemic attack (TIA), cerebral hemorrhage and transient neurological deficit) and death or dependent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who diagnosed with moyamoya disease
2. Adults 18 to 65 years of age
3. The onset symptoms manifested as ischemic symptoms (TIA or stroke) or atypical symptoms (headache, epilepsy or asymptomatic)
4. Able to receive the necessary imaging examination
5. Patients who pre-agreed to the study

Exclusion Criteria:

1. Prior cerebral hemorrhage history
2. Other brain or cerebrovascular disease
3. Previous history of revascularization surgery
4. Dependent (mRS > 2)
5. Receive other type of revascularization surgery
6. Peripheral blood vessel disease (especially subclavian arterial and upper limb artery stenosis or occlusion).
7. Patients who do not agree with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With Cerebrovascular Events. | postoperative one month
  Cerebrovascular events included ischemic stroke, transient ischemic attack (TIA), cerebral hemorrhage and hyperperfusion syndrome.
Number of Patients Dependent or Death | postoperative one month
  Dependent included the modified Rankin Scale (mRS) > 2. Death included any reason caused death.

SECONDARY OUTCOMES:
The Severity of the Ischemic Stroke after Surgery | postoperative one month
  The severity of the ischemic stroke was evaluated by the white matter hyperintensities volume on the MRI, the neurological deficits duration and the Modified Rankin Scale (mRS) of patients.
Number of Patients Occured Re-stroke at Follow-up Period | 6 months and 12 months after EDAS
  Re-stroke included ischemic stroke and hemorrhagic stroke.
Number of Patients Dependent or Death at Follow-up Period | 6 months and 12 months after EDAS
  Dependent included the modified Rankin Scale (mRS) > 2. Death included any reason caused death.
Number of Patients with Improved Neurological Function at Follow-up Period | 6 months and 12 months after EDAS
  The modified Rankin Scale (mRS) decreased at the follow-up period compared to preoperative scores
Perfusion Status of Patients at Follow-up Period | 6 months and 12 months after EDAS
  The perfusion status detected by stages of pre-infarction period based on computed tomography perfusion imaging
Number of Patients With Any Side Effects of Remote Ischemic Preconditioning (RIPC) Treatment. | From baseline to 12 months after treatment
  The side effects referred to any side effects of RIPC or sham RIPC treatment, not including the sides effect of medications and EDAS.
Participants Who Got New Diffusion-weighted Imaging (DWI) Lesions on Post-treatment Magnetic Resonance Imaging (MRI) Scans. | Within 48 hours after EDAS
  The presence of ≥1 new brain lesions on DWI

CONTACTS AND LOCATIONS:
Overall Officials: Yuanli Zhao, MD, Principal Investigator — Beijing Tiantan Hospital; Rong Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hosiptal, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) of this study are available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after the study ended
Access Criteria: The IPD of this study are available from the principal investigator upon reasonable request.

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250